CLINICAL TRIAL: NCT05486169
Title: Gastroesophageal Reflux Disease in Patients Before and After Laparoscopic Sleeve Gastrectomy - pH-impedance Monitoring
Brief Title: Gastroesophageal Reflux Disease After Laparoscopic Sleeve Gastrectomy
Acronym: SLEEFLUX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warmia and Mazury in Olsztyn (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Natalia Dowgiałło-Gornowicz, MD, PhD, assistant professor, University of Warmia and Mazury in Olsztyn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2022/06/X/NZ5/00007
Record Dates: First submitted 2022-07-30; First posted 2022-08-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Gastroesophageal Reflux; Obesity
Keywords: Gastroesophageal Reflux Disease; GERD; Obesity Surgery; Sleeve gastrectomy
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sleeve Gastrectomy — surgery of laparoscopic sleeve gastrectomy

SUMMARY:
The planned research is to analyze the occurrence of gastroesophageal reflux disease (GERD) before and after sleeve gastrectomy (SG). The study includes patients with BMI above 40 kg / m2 without symptoms of GERD before surgery and any pathological changes in gastroscopy. The day before the surgery, patients will be tested with impedance pH measurement. Thereafter, patients will undergo SG according to standard technique. As part of the follow-up 6 months after the surgery, the pH-measurement test with impedance again will be performed again for evaluation of the occurrence of GERD after surgery. It was planned to include 50 people in the study.

The main aim of the study is to assess the frequency and quality of GERD in patients after SG.

DETAILED DESCRIPTION:
According to World Health Organization data, almost 15% of people in the world are obese, and this is constantly growing. According to the available literature, an effective method of observation long-term treatment that allows for the permanent cure of obesity is surgical treatment. Currently sleeve gastrectomy (SG) is the most commonly performed procedure in the world. There are numerous evidence of the effectiveness of surgery in treating obesity and comorbidities, however, came along with the increase in the number of procedures performed, controversy arises, including the occurrence of gastroesophageal reflux disease (GERD) after surgery. As a consequence, GERD can lead to esophageal cancer. This problem wants to be dealt with in this study.

The planned research is to analyze the occurrence of GERD before and after SG. Down the study will include patients whose BMI is 40 kg / m2 and more who will be positive passed the qualification process for SG. The exclusion criteria are the occurrence of symptoms of GERD before surgery, pathological changes in gastroscopy - features of reflux oesophagitis, and the patient's lack of consent to participation in the study. On the eve of surgery, patients will be tested with impedance pH measurement. Is it non-invasive 24-hour examination consisting in measuring the pH and impedance of the esophagus allowing for the detection of reflux episodes and their accurate assessment - type, time. Currently this test is the gold standard for the diagnosis of GERD, including in patients asymptomatic. Thereafter, patients will undergo SG according to standard technique. As part of the follow-up 6 months after the surgery, the pH-measurement test with impedance again will be performed again for evaluation of the occurrence of GERD after surgery. It was planned to include 50 people in the study, which is good, satisfactory material for statistical analysis.

The main aim of the study is to assess the frequency and quality of GERD in patients after SG. Yet published works on this issue define the occurrence of GERD mainly on on the basis of an interview with the patient or changes in the gastroscopy examination, which does not allow definitive definition of the disease incidence. Often, the mileage may be left to the patient asymptomatic - e.g. in the case of neutral reflux, and changes in endoscopic examination may not yet be visible. Thus, the only effective method to assess the occurrence of GERD is to perform a pH-measurement test with impedance. Moreover a group of 50 people subjected to the tests will make it possible to try to determine the predisposing factors to the occurrence of GERD after surgery, which will enable further the order of taking actions to prevent its occurrence. The results of the research will be presented on a thematic basis scientific conferences, then published in one of the renowned journals research in this field.

ELIGIBILITY:
Inclusion Criteria:

* BMI above 40kg/m2
* positive qualification process for laparoscopic sleeve gastrectomy

Exclusion Criteria:

* symptoms of gastroesophageal reflux disease before the surgery
* pathological changes in gastroscopy before the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
gastroesophageal reflux after sleeve gastrectomy | 6 months
  The main aim of the study is to assess the frequency and quality of gastroesophageal reflux disease in patients six months after sleeve gastrectomy. The reflux will be measured in each patient using 24-hour pH-impedance testing

SECONDARY OUTCOMES:
outcomes of sleeve gastrectomy | 6 months
  Each patient would have their body weight measured and asked about the resolution of comorbidities during the control visit six months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- UWM, Olsztyn, Poland

IPD SHARING:
Plan to Share IPD: No